CLINICAL TRIAL: NCT04901260
Title: AMAZE™ Asthma Implementation Quality Improvement Study
Brief Title: AMAZE™ Asthma Implementation QI Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Greater Austin Allergy (Unknown); Evidera, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: N3566000000
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Quality Initiative: Each participant will be asked to complete the symptoms log daily for up to 6 months. Additional surveys will be completed throughout the study by participants and GAA clinical staff.
  Interventions: Device: AMAZE™ Disease Management Platform

INTERVENTIONS:
Device: AMAZE™ Disease Management Platform — The disease management platform includes a patient mobile application where patients can enter daily symptoms, communicate with their healthcare providers, and access educational materials. Additionally, the healthcare providers will have access to a dashboard that is integrated with the EMR and patient app.

SUMMARY:
The primary study objective is to generate evidence as to the feasibility, usability, perceived value, and potential benefits of implementing the AMAZE™ platform into clinical practice.

DETAILED DESCRIPTION:
AstraZeneca has developed the AMAZE™ disease management platform to be used across multiple disease indications to provide a unified experience for the management of patients throughout their patient care journey. AMAZE™ integrates multiple systems, including a patient mobile application where patients can enter daily symptoms and impact to communicate this information to their healthcare provider, as well as access disease educational materials. Implementation of AMAZE™ within clinical practice has not yet been evaluated. The results from this study will be used to inform any changes or modifications that need to be made to the technology platform, its implementation process, and explore impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age at the time of enrollment
* Clinically confirmed diagnosis of asthma
* Access to a smartphone with internet access with the following requirements: iOS (Operating System iOS 13 or newer and Devices iPhone 8 or newer) or Android (Operating System 8.0 or newer)
* Able to understand and speak English sufficiently to be able to use the AMAZE™ patient App
* Willingness to participate in a telephone interview and be audio-recorded
* Consenting to participate in the study

Exclusion Criteria:

* Current diagnosis of active chronic obstructive pulmonary disease (COPD) or any pulmonary diagnosis other than asthma;
* Has a cognitive impairment, hearing difficulty, acute psychopathology, medical condition, or insufficient knowledge of the English language that, in the opinion of the investigator, would interfere with his or her ability to agree to participate and/or complete the ACT™

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the GAA network, with approximately 120 patients ≥18 years old with a current diagnosis of asthma being enrolled. Participants will need to have access to a smartphone with internet.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Patient App Usage | Up to 6 months
  Patient app usage will be measured as the number of days the patient engages (i.e., completes daily log, sends a message) with the app at least once a day during the study period.
Clinician Dashboard Usage | Up to 6 months
  Clinician dashboard usage will be measured as the mean number of days per week/month that the clinical site staff accessed the AMAZE™ dashboard over the 6-month period.
Daily Asthma status | Up to 6 months
  Patient daily asthma status (bad, okay, good) reported on the app will be described weekly during Month 1, and then per month from Month 1 through Month 6 pending availability of data after Month 1.
Symptoms and Triggers | Up to 6 months
  Frequency of symptoms and frequency of triggers (for those that reported symptoms) reported on the app will be described weekly during Months 1, and then per month from Month 1 through Month 6 pending availability of data after Month 1.
Self-Reported Rescue Medication usage | Up to 6 months
  The number of times per month a patient used rescue medication as well as visited the emergency room or urgent care as reported on the app will be described from Month 1 through Month 6.

SECONDARY OUTCOMES:
Impact of AMAZE™ on patient visits | Up to 6 months
  The impact of AMAZE™ on patient visits will be measured as the frequency of patients who select "agree" or "strongly agree" in response to the 9-items in the patient visit experience survey.
ER visits and Hospitalization avoidance | Up to 6 months
  The impact of AMAZE™ on ER and hospitalizations will be measured as the frequency of patients who report "agree" or "strongly agree" with the item "The visit helped avoid an ER or Urgent Care center visit or hospitalization" from the patient visit experience survey
Patient Perception of Appointment Discussions and Taking Part in Asthma Decisions | Up to 6 months
  The impact of AMAZE™ on improved patient communication with their provider will be measured as the frequency of patients who report "agree" or "strongly agree" with the items "the app helped me discuss my asthma with my healthcare provider(s) during my most recent visit" and "I was included in making decisions about my asthma treatment during my most recent visit" on the patient visit experience survey.
Patient Perception of Usability and Design of Mobile app | Up to 6 months
  The usability of the AMAZE™ app will be measured by the frequency of patients who rate the app excellent (SUS score >80.3), good (68-80.3), okay (68), poor (51-68), or awful (<51) at months 1 and 6
Clinical Staff Perception of Usability and Design of Dashboard | Up to 6 months
  The usability of the AMAZE™ dashboard will be measured by the frequency of clinical staff who rate the app excellent (SUS score >80.3), good (68-80.3), okay (68), poor (51-68), or awful (<51) at months 1 and 6
Evaluate ease of implementation of AMAZE™ in clinical setting | Up to 6 months
  The ease of implementation of AMAZE™ will be measured by the frequency of clinical staff who report "very easy" or "somewhat easy" to the question "How would you rate the overall ease of implementing AMAZE™ on a platform into your clinical practice?" in the post-study survey at month 6.
Evaluate impact of AMAZE™ on managing patients | Up to 6 months
  The impact of AMAZE™ on managing patients will be measured by the frequency of clinical staff who report "moderately" or "very well" to the question "Did the AMAZE™ help you manage your patients?" in the post-study survey at month 6.
Evaluate Perceived Benefit of AMAZE™ in clinical setting | Up to 6 months
  The perceived benefit of AMAZE™ will be evaluated by the frequency of clinical staff who endorse different perceived benefits based on the item "what did you find the most useful about the AMAZE™ platform?" in the post-study survey at month 6.
Evaluate Perceived Disadvantages of AMAZE™ in clinical setting | Up to 6 months
  The perceived disadvantages of AMAZE™ will be evaluated by the frequency of clinical staff who endorse different perceived disadvantages based on the item "what did you find the least useful or cumbersome about the AMAZE™ platform?" in the post-study survey at month 6.
Evaluate patient satisfaction with healthcare experience | Up to 6 months
  Patient satisfaction with their healthcare experience will be evaluated using the PSQ-18 items and subscale scores (General Satisfaction, Technical Quality, Interpersonal Manner, Communication, Financial Aspects, Time Spent with Doctor, Accessibility and Convenience) at Month 6.
Evaluate patient satisfaction with app | Up to 6 months
  Satisfaction with the app features will be measured by the frequency of patients who report satisfaction on a scale of 1 (lowest satisfaction) to 5 (highest satisfaction) at months 1, 3, and 6.

OTHER OUTCOMES:
Evaluating change in medication | Up to 6 months
  Medication changes from baseline to six-month will be evaluated.
Evaluating clinician-reported asthma control | Up to 6 months
  Asthma control was assessed by a clinician completed single item; asthma control at baseline will be evaluated.
Evaluating patient-reported asthma control | Up to 6 months
  The impact of AMAZE™ on asthma control will be measured as the frequency of patients considered to be poorly controlled (ACT scores ≤15), not well-controlled (ACT scores 16-19, and well-controlled (ACT scores ≥20) from Month 1 through Month 6.
Changes in asthma symptoms before clinical visit | Up to 6 months
  Frequency of symptoms reported in the patient daily log up to a week proceeding a clinical visit during the study period will be evaluated to assess trends in symptoms that may have triggered a visit.
Changes in medication after clinical visit | Up to 6 months
  Following a clinical visit any time during the study period, medication changes will be monitored to determine if any changes were prompted by the visit.
Characteristics of Patients Most Likely to Benefit from AMAZE™ | Up to 6 months
  Demographic information reported by the patient and clinical information reported by the clinical staff will be used and stratified by subgroups, including age, asthma severity, education, and ethnicity, to evaluate characteristics of patients most likely to benefit from AMAZE™

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schultz, DO, MPH, Principal Investigator — GAA
Locations (1):
- Research Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Alladina J, Moschovis PP, Gandhi HN, Carstens D, Bacci ED, Cutts K, Coyne KS, Goldsborough K, Jiang D, O'Brien C, Bernard Kinane T. Observational study of the Amaze asthma disease management platform. Digit Health. 2024 Oct 22;10:20552076241282380. doi: 10.1177/20552076241282380. eCollection 2024 Jan-Dec. PMID 39479373
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=N3566000000&attachmentIdentifier=80d573a4-d884-4b40-b467-bf59934f923c&fileName=EVA-28838_AMAZE_Redacted_Synopsis_20July2022_Clean_V2.pdf&versionIdentifier=